CLINICAL TRIAL: NCT05995951
Title: Deep Brain Stimulation Surgery for the Treatment of Refractory Obsessive-Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Idit tamit, Principal Investigator, Rabin Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1005-20-RMC
Record Dates: First submitted 2023-04-17; First posted 2023-08-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Bran Stimulation (DBS) - Treatment group (Other): Treatment group will undergo Deep Bran Stimulation (DBS) for OCD (targeting the amSTN) for four months.
  At the end of four months treatment, the groups will be crossed-over for another four months. Thus, the sham group will start active stimulation and the treatment group will start sham treatment for four months.
  Interventions: Device: Deep Bran Stimulation (DBS)
- Sham-control (Other): sham stimulation for four months.
  At the end of four months treatment, the groups will be crossed-over for another fourmonths. Thus, the sham group will start active stimulation and the treatment group will start sham treatment for four months.
  Interventions: Device: Sham-stimulation

INTERVENTIONS:
Device: Deep Bran Stimulation (DBS) — Deep brain stimulation (DBS) surgery targeting the antero-medial Sub-Thalamic Nucleus (amSTN)
  Arms: Deep Bran Stimulation (DBS) - Treatment group
Device: Sham-stimulation — Deep brain stimulation (DBS) surgery - Sham stimulation
  Arms: Sham-control

SUMMARY:
This study will include two parts. The first part will include two patients in a non-blinded, non-randomized, open trial. They will undergo Deep Bran Stimulation (DBS) for OCD (targeting the amSTN), as clinically accepted and approved in Israel (by the MOH) and in other countries in Europe and the US. The second part will include eight patients. This part will be an interventional, randomized, double-blinded clinical trial (patient and psychiatrist; the neurosurgeon will activate stimulation during the randomization period and will not be blinded). All subjects will undergo standard pre-operative psychiatric and neurosurgical assessment. Around 4-6 weeks later subjects will undergo implantation of Medtronic implantable DBS system (bilateral brain leads model 3389, lead extenders and PERCEPT pulse generator). Intraoperative recordings will include single unit and local field potentials (LFP) for target identification and validation, as accepted for clinical use. In the second part of the study, blinded randomization for treatment or sham-control arms (1:1 ratio) will be held two weeks post-operation. Treatment and sham-control arms will continue for four months. At the end of four months treatment, the groups will be crossed-over for another four months. Thus, the sham-control group will start treatment (using pre-defined stimulation parameters) and the treatment group will start sham stimulation. Four months later (six and a half months from surgery), randomization will be over, and both arms will get open-label active treatment. Psychiatric assessments post-operation will take place after two weeks, one month, and then once every six weeks, in the first year for all study patients. Chronic recordings will take place using the clinically used and approved PERCEPT DBS pulse generator during the first year after surgery.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is characterized by the presence of intrusive obsessions, compulsions, or both. Despite undergoing optimal pharmacological and psychological treatment, around a tenth of patients remain with refractory OCD, with a great impact on their everyday function and quality of life.

Deep brain stimulation (DBS) surgery is a safe and effective treatment, used for movement disorders for over 20 years now, and lately was approved worldwide also for intractable epilepsy. In the past decade, many studies of DBS for refractory OCD proved safety and effectiveness with 50% reduction in OCD symptoms of the most refractory patients.

This study will include two parts. The first part will include two patients in a non-blinded, non-randomized, open trial. They will undergo Deep Bran Stimulation (DBS) for OCD (targeting the amSTN), as clinically accepted and approved in Israel (by the MOH) and in other countries in Europe and the US. The second part will include eight patients. This part will be an interventional, randomized, double-blinded clinical trial (patient and psychiatrist; the neurosurgeon will activate stimulation during the randomization period and will not be blinded). All subjects will undergo standard pre-operative psychiatric and neurosurgical assessment. Around 4-6 weeks later subjects will undergo implantation of Medtronic implantable DBS system (bilateral brain leads model 3389, lead extenders and PERCEPT pulse generator). Intraoperative recordings will include single unit and local field potentials (LFP) for target identification and validation, as accepted for clinical use. In the second part of the study, blinded randomization for treatment or sham-control arms (1:1 ratio) will be held two weeks post-operation. Treatment and sham-control arms will continue for four months. At the end of four months treatment, the groups will be crossed-over for another four months. Thus, the sham-control group will start treatment (using pre-defined stimulation parameters) and the treatment group will start sham stimulation. four months later (six and a half months from surgery), randomization will be over, and both arms will get open-label active treatment. Psychiatric assessments post-operation will take place after two weeks, one month, and then once every six weeks, in the first year for all study patients. Chronic recordings will take place using the clinically used and approved PERCEPT DBS pulse generator during the first year after surgery.

Primary aims:

1. Assess the effects of the anteromedial sub-thalamic nucleus (amSTN)/medial forebrain bundle (MFB) stimulation on obsessive/compulsive symptoms
2. Map the amSTN using neuronal responses (single unit and LFP recordings) to cognitive-emotion provocation task during surgery
3. Record chronic brain activity with the implanted pulse generator and look for neuronal signatures correlated with symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of obsessive-compulsive disorder according to DSM 5 criteria, diagnosed by three independent psychiatrists not routinely involved with the patients' treatment.
* Severe OCD assessed by the Yale-Brown Obsessive-Compulsive Scale (YBOCS) with a score of more than 25.
* Refractory OCD; severe symptoms and impairment for more than 5 years despite pharmacological and psychological treatment.
* Have failed to improve following treatment with at least two serotonin transport inhibitors and one augmenting agent taken for an adequate time period.
* Having failed to improve despite adequate psychotherapy.
* Meet established criteria for implantation of a deep brain stimulation system.
* Patients between ages 18 and 75.
* Ability to understand and sign written informed consent by the patient.

Exclusion Criteria:

* Diagnosis of severe major depression disorder (MDD) with psychotic features.
* Significant suicidal risk [Hamilton Depression scale item 3 (suicide) >2].
* Comorbidity with any primary Psychotic Disorder, Bipolar Disorder, Post-Traumatic Stress Disorder (PTSD), Eating Disorder, Autistics Spectrum Disorder.
* History of substance or alcohol dependence or abuse in the preceding 12 months.
* Significant cognitive decline, measured by Mini-Mental State Examination (MMSE <26) and Montreal Cognitive Assessment (MoCA; <24).
* Any other current clinically significant neurological disorder or medical illness affecting brain function, other than a tic disorder.
* Any clinically significant abnormality on preoperative MRI.
* Any DBS contraindication, infection, coagulopathy, significant cardiac risk factors, or other significant medical risk factors for surgery.
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms - YBOCS score (0-40) | baseline (before stimulation initiation)
  Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms. This will be assessed by the YBOCS. More than a 35% reduction on the YBOCS will be considered clinically significant. YBOCS score (0-40) - lower scores mean a better outcome.
Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms - YBOCS score (0-40) | four months post-implantation
  Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms. This will be assessed by the YBOCS. More than a 35% reduction on the YBOCS will be considered clinically significant. YBOCS score (0-40) - lower scores mean a better outcome.
Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms - YBOCS score (0-40) | eight months post-implantation
  Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms. This will be assessed by the YBOCS. More than a 35% reduction on the YBOCS will be considered clinically significant. YBOCS score (0-40) - lower scores mean a better outcome.
Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms - YBOCS score (0-40) | 12 months post-implantation
  Assessment of the efficacy of amSTN/MFB stimulation on OCD symptoms. This will be assessed by the YBOCS. More than a 35% reduction on the YBOCS will be considered clinically significant. YBOCS score (0-40) - lower scores mean a better outcome.
Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures | baseline (before stimulation initiation)
  Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures. This will be measured by correlating various measures of discharge (rate, amplitude, coherence, phase, burstiness, and cross-frequency coupling) and task-related activity (magnitude of modulation, directionality, and amplitude sensitivity) with the severity of cognitive and mood impairments of patients undergoing surgery.
Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures | four months post-implantation
  Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures. This will be measured by correlating various measures of discharge (rate, amplitude, coherence, phase, burstiness, and cross-frequency coupling) and task-related activity (magnitude of modulation, directionality, and amplitude sensitivity) with the severity of cognitive and mood impairments of patients undergoing surgery.
Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures | eight months post-implantation
  Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures. This will be measured by correlating various measures of discharge (rate, amplitude, coherence, phase, burstiness, and cross-frequency coupling) and task-related activity (magnitude of modulation, directionality, and amplitude sensitivity) with the severity of cognitive and mood impairments of patients undergoing surgery.
Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures | 12 months post-implantation
  Assessment of the association between amSTN electrophysiological discharge and cognitive/ emotional measures. This will be measured by correlating various measures of discharge (rate, amplitude, coherence, phase, burstiness, and cross-frequency coupling) and task-related activity (magnitude of modulation, directionality, and amplitude sensitivity) with the severity of cognitive and mood impairments of patients undergoing surgery.

SECONDARY OUTCOMES:
The effects of DBS on mood | baseline (before stimulation initiation)
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).
The effects of DBS on mood | four months post-implantation
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).
The effects of DBS on mood | eight months post-implantation
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).
The effects of DBS on mood | 12 months post-implantation
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).
The effects of DBS on quality of life | baseline (before stimulation initiation)
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).
The effects of DBS on quality of life | four months post-implantation
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).
The effects of DBS on quality of life | eight months post-implantation
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).
The effects of DBS on quality of life | 12 months post-implantation
  The effects of DBS on mood and quality of life will be tested using various scales: Hamilton Scale for Anxiety (HAM-A), Hamilton Scale for Depression (HAM-D21), Brief Psychiatric Rating Scale (BPRS), overall state (Clinical Global Inventory [CGI]), and Mini-Mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Overall Officials: Idit Idit, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided